CLINICAL TRIAL: NCT05468320
Title: An Open-label, Single-arm, Multicenter Study to Evaluate the Efficacy and Safety of Caplacizumab and Immunosuppressive Therapy Without Firstline Therapeutic Plasma Exchange in Adults With Immune-mediated Thrombotic Thrombocytopenic Purpura
Brief Title: Caplacizumab and Immunosuppressive Therapy Without Firstline Therapeutic Plasma Exchange in Adults With Immune-mediated Thrombotic Thrombocytopenic Purpura
Acronym: MAYARI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFC16521; U1111-1244-0426 (Registry Identifier: ICTRP); 2024-513262-19 (Registry Identifier: CTIS); 2022-001177-31 (EudraCT Number)
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Thrombotic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — caplacizumab; Adrenal Cortex Hormones; Prednisone; Prednisolone; Rituximab; Biosimilar Pharmaceuticals

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Caplacizumab & immunosuppressive therapy without 1st-line TPE (Experimental): All participants will receive open label caplacizumab daily and immunosuppressive therapy (corticosteroid +/-anti-CD20 therapy antibody [rituximab or biosimilar]) without first line TPE
  Interventions: Drug: Caplacizumab; Drug: Corticosteroids; Biological: anti-CD20 antibody

INTERVENTIONS:
Drug: Caplacizumab — Lyophilized powder for solution for injection.
  Other Names: Cablivi®
Drug: Corticosteroids — Solution for injection or Tablet
  Other Names: Prednisone® /Prednisolone®
Biological: anti-CD20 antibody — Solution for injection
  Other Names: rituximab or biosimilar

SUMMARY:
This is a single group, treatment, Phase 3, open-label, single-arm study to evaluate the efficacy and safety of caplacizumab and immunosuppressive therapy (IST) without firstline therapeutic plasma exchange (TPE) with primary endpoint of remission in male and female participants aged 18 to 80 years with immune-mediated thrombotic thrombocytopenic purpura (iTTP).

The anticipated study duration per participant without a recurrence while on therapy is maximum 24 weeks (ie, approximately 1 day for screening + maximum 12 weeks of treatment for the presenting episode + 12 weeks of follow-up). Participants will have daily assessments during hospitalization and weekly visits for assessments during ongoing treatment with caplacizumab and IST. There will be 3 outpatient visits for assessments during the follow-up period. There will be two additional follow-up visits for participants who do not have ADAMTS13 activity levels of ≥50% at the time of caplacizumab discontinuation.

DETAILED DESCRIPTION:
The anticipated study duration per participant with the presenting episode therefore is a maximum of about 24 weeks (ie, 1 day of screening + maximum 12 weeks of treatment for the presenting episode + 12 weeks of follow-up).

ELIGIBILITY:
Inclusion Criteria:

Participants with a clinical diagnosis of iTTP (initial or recurrent), which includes thrombocytopenia, microangiopathic hemolytic anemia (eg, presence of schistocytes in peripheral blood smear) and relatively preserved renal function. The iTTP diagnosis should be confirmed by ADAMTS13 testing within 48 hours (2 days).

Participants with a clinical diagnosis of iTTP and a French TMA score of 1 or 2.

A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

* Is a woman of nonchildbearing potential (WONCBP), OR
* Is a woman of childbearing potential (WOCBP) and agrees to use an acceptable contraceptive method during the overall treatment period and for at least 2 months after the last study drug administration.

Male participants with female partners of childbearing potential must agree to follow the contraceptive guidance as per protocol during the overall treatment period and for at least 2 months after last study drug administration.

Exclusion Criteria:

Platelet count ≥100 x 10^9/L. Serum creatinine level >2.26 mg/dL (200 µmol/L) in case platelet count is >30 x 10^9/L (to exclude possible cases of atypical HUS).

Known other causes of thrombocytopenia including but not limited to:

* Clinical evidence of enteric infection with E. coli 0157 or related organism.
* Atypical HUS.
* Hematopoietic stem cell, bone marrow or solid organ transplantation-associated thrombotic microangiopathy.
* Known or suspected sepsis.
* Diagnosis of disseminated intravascular coagulation. Congenital TTP (known at the time of study entry). Clinically significant active bleeding or known co-morbidities associated with high risk of bleeding (excluding thrombocytopenia).

Inherited or acquired coagulation disorders. Malignant arterial hypertension. Participants requiring or expected to require invasive procedures immediately (eg, stroke requiring thrombolytic therapy, those who need mechanical ventilation, etc.).

Those presenting with severe neurological or cardiac disease. Clinical condition other than that associated with TTP, with life expectancy <6 months, such as end-stage malignancy.

Known chronic treatment with anticoagulants and anti-platelet drugs that cannot be stopped (interrupted) safely, including but not limited to:

* vitamin K antagonists.
* direct-acting oral anticoagulants.
* heparin or low molecular weight heparin (LMWH).
* non-steroidal anti-inflammatory molecules other than acetyl salicylic acid. Participants who were previously enrolled in this clinical study (study EFC16521).

Participants who received an investigational drug, or device, other than caplacizumab, within 30 days of anticipated IMP administration or 5 half-lives of the previous investigational drug, whichever is longer.

Positive result on COVID test.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2024-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (27):
- United States (4):
  - University of Alabama- Site Number : 8400011, Birmingham, Alabama
  - Johns Hopkins University- Site Number : 8400007, Baltimore, Maryland
  - Duke University Medical Center Site Number : 8400022, Durham, North Carolina
  - The Ohio State University Comprehensive Cancer Center - Site Number : 8400001, Columbus, Ohio
- Investigational Site Number : 0560003, Yvoir, Belgium
- Investigational Site Number : 1240001, Toronto, Ontario, Canada
- Czechia (2):
  - Investigational Site Number : 2030001, Brno
  - Investigational Site Number : 2030003, Prague
- France (4):
  - Investigational Site Number : 2500002, Bois-Guillaume
  - Investigational Site Number : 2500005, Lille
  - Investigational Site Number : 2500003, Paris
  - Investigational Site Number : 2500001, Paris
- Germany (4):
  - Investigational Site Number : 2760006, Berlin
  - Investigational Site Number : 2760002, Cologne
  - Investigational Site Number : 2760001, Frankfurt am Main
  - Investigational Site Number : 2760004, Hanover
- Italy (5):
  - Investigational Site Number : 3800003, Avellino, Campania
  - Investigational Site Number : 3800001, Milan, Lombardy
  - Investigational Site Number : 3800006, Genova
  - Investigational Site Number : 3800005, Verona
  - Investigational Site Number : 3800004, Vicenza
- Japan (2):
  - Investigational Site Number : 3920003, Kurashiki-shi, Okayama-ken
  - Investigational Site Number : 3920001, Iruma-gun, Saitama
- Investigational Site Number : 5280002, Amersfoort, Netherlands
- Investigational Site Number : 7240001, Madrid / Madrid, Madrid, Comunidad de, Spain
- United Kingdom (2):
  - Investigational Site Number : 8260001, London, London, City of
  - Investigational Site Number : 8260002, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Volker LA, Brinkkotter PT. Tailored treatment of acute immune-mediated thrombotic thrombocytopenic purpura. Hematology Am Soc Hematol Educ Program. 2025 Dec 5;2025(1):614-620. doi: 10.1182/hematology.2025000757. PMID 41348038
- See also: EFC16521 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25249&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 27 centers in 11 countries. A total of 58 participants were screened between 21 November 2022 and 24 June 2024, of which 2 were screen failures, and 5 participants treated with at least 1 dose of caplacizumab were not enrolled due to not meeting study eligibility criteria.
Pre-assignment Details: A total of 51 participants were enrolled in the study.
Groups:
- Caplacizumab and IST Without First-Line TPE: Participants received open-label caplacizumab daily and immunosuppressive therapy (IST) (corticosteroid +/-anti-CD20 antibodies [Ab] therapy [rituximab or biosimilar]) without first-line therapeutic plasma exchange (TPE). Participant received caplacizumab 10 milligram (mg) intravenous (IV) injection for a single dose followed by caplacizumab 10 mg subcutaneous (SC) injection 4 to 6 hours after the IV dose on Day 1. Then participants received caplacizumab 10 mg SC injection daily starting on Day 2 for a maximum treatment duration of 12 weeks. Participants also received corticosteroids (prednisone or prednisolone) 1 to 1.5 mg/kilogram (kg)/day, IV or oral for 1 week and taper over 3 to 4 weeks, along with anti-CD20 Ab therapy at the beginning of the study. Participants did not receive TPE as first-line therapy, however, they could receive TPE if it was determined that there was a lack of adequate response to study treatment or if there was any clinical deterioration at any time during the study, including during the first 24 hours.
Period: Overall Study
Arm/Group | Caplacizumab and IST Without First-Line TPE
Started | 51
Completed | 49
Not Completed | 2
Not completed — Other | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: The enrolled population consisted of all participants from the screened population who met the eligibility criteria.
Groups:
- Caplacizumab and IST Without First-Line TPE: Participants received open-label caplacizumab daily and IST (corticosteroid +/-anti-CD20 Ab therapy [rituximab or biosimilar]) without first-line TPE. Participant received caplacizumab 10 mg IV injection for a single dose followed by caplacizumab 10 mg SC injection 4 to 6 hours after the IV dose on Day 1. Then participants received caplacizumab 10 mg SC injection daily starting on Day 2 for a maximum treatment duration of 12 weeks. Participants also received corticosteroids (prednisone or prednisolone) 1 to 1.5 mg/kg/day, IV or oral for 1 week and taper over 3 to 4 weeks, along with anti-CD20 Ab therapy at the beginning of the study. Participants did not receive TPE as first-line therapy, however, they could receive TPE if it was determined that there was a lack of adequate response to study treatment or if there was any clinical deterioration at any time during the study, including during the first 24 hours.
Arm/Group | Caplacizumab and IST Without First-Line TPE
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 8
  White | 20
  More than one race | 0
  Unknown or Not Reported | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Remission Without Requirement of Therapeutic Plasma Exchange During Overall Study Period
Description: Remission was defined as sustained clinical response with either no TPE and no anti- von Willebrand factor (vWF) therapy for >=30 days (clinical remission) or with attainment of a disintegrin and metalloproteinase with a thrombospondin type 1 motif13 (ADAMTS13) activity level >=50% (complete ADAMTS13 remission), whichever occurred first. Clinical response was defined as sustained platelet count >=150 × 10^9/liter (L) and lactate dehydrogenase (LDH) <1.5 × upper limit of normal (ULN) and no clinical evidence of new or progressive ischemic organ injury for at least 2 consecutive visits.
Time Frame: From first dose of study treatment (Day 1) up to end of follow-up (up to approximately 24 weeks)
Population: The modified intent-to-treat (mITT) population consisted of all enrolled participants who received at least 1 dose of the study treatment with an evaluable primary endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Caplacizumab and IST Without First-Line TPE
Number analyzed (Participants) | 46
percentage of participants | 93.5 [82.5 to 97.8]

2. Secondary Outcome: Percentage of Participants Who Achieved Remission During Overall Study Period
Description: Remission was defined as sustained clinical response with either no TPE and no anti- vWF therapy for >=30 days (clinical remission) or with ADAMTS13 activity level >=50% (complete ADAMTS13 remission), whichever occurred first. Clinical response was defined as sustained platelet count >=150 × 10^9/L and LDH <1.5 × ULN and no clinical evidence of new or progressive ischemic organ injury for at least 2 consecutive visits.
Time Frame: From first dose of study treatment (Day 1) up to end of follow-up (up to approximately 24 weeks)
Population: The mITT population consisted of all enrolled participants who received at least 1 dose of the study treatment with an evaluable primary endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Caplacizumab and IST Without First-Line TPE
Number analyzed (Participants) | 46
percentage of participants | 95.7 [85.5 to 98.8]

3. Secondary Outcome: Percentage of Participants Who Required Therapeutic Plasma Exchange During On-Treatment Period
Description: TPE was a procedure in which blood of the participant was passed through a medical device which separated out plasma from other components of blood and the participant's plasma was removed and replaced with a replacement solution such as colloid solution (example, albumin and/or plasma) or a combination of crystalloid/colloid solution. TPE replenishes the ADAMTS13 enzyme and removes anti-ADAMTS13 antibodies, and ultra-large von Willebrand factor multimers gradually from the circulation.
Time Frame: From first dose of study treatment (Day 1) up to last dose of study treatment, approximately 12 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Caplacizumab and IST Without First-Line TPE
Number analyzed (Participants) | 46
percentage of participants | 4.3 [1.2 to 14.5]

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (TESAEs), and Treatment-Emergent Adverse Events of Special Interest (TEAESI)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. TEAEs were defined as the AEs that developed, worsened or became serious during the treatment-emergent period. SAE: Any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or was a congenital anomaly/birth defect, or any other situation where medical or scientific judgment of investigator were exercised. An AESI is an AE (serious or nonserious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor was required.
Time Frame: From first dose of study treatment (Day 1) up to last dose of study treatment + 28 days (approximately 16 weeks)
Population: The safety population consisted of all enrolled participants who took at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Caplacizumab and IST Without First-Line TPE
Number analyzed (Participants) | 50
Participants
  TEAEs | 46
  TESAEs | 7
  TEAESI | 8

5. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response During On-Treatment Period
Description: Clinical response was defined as sustained platelet count >=150 × 10^9/L and LDH <1.5 × ULN and no clinical evidence of new or progressive ischemic organ injury for at least 2 consecutive visits.
Time Frame: From first dose of study treatment (Day 1) up to last dose of study treatment, approximately 12 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Caplacizumab and IST Without First-Line TPE
Number analyzed (Participants) | 46
percentage of participants | 97.8 [88.7 to 99.6]

6. Secondary Outcome: Percentage of Participants Who Achieved Clinical Response During Overall Study Period
Description: as for outcome 5
Time Frame: From first dose of study treatment (Day 1) up to end of follow-up (up to approximately 24 weeks)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Caplacizumab and IST Without First-Line TPE
Number analyzed (Participants) | 46
percentage of participants | 97.8 [88.7 to 99.6]

7. Secondary Outcome: Time to Platelet Count Response
Description: Time to platelet count response was defined as time from start of study treatment to initial platelet count >=150 × 10^9/L that was sustained for >=2 days.
Time Frame: From first dose of study treatment (Day 1) up to end of follow-up (up to approximately 24 weeks)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Caplacizumab and IST Without First-Line TPE
Number analyzed (Participants) | 46
days | 4 [3 to 5]

8. Secondary Outcome: Percentage of Participants Refractory to Therapy During On-Treatment Period
Description: Refractory to therapy was defined as lack of sustained platelet count increment (over 2 consecutive days) or platelet counts <50 × 10^9/L and persistently elevated LDH (>1.5 × ULN) despite 5 days of treatment during the on-treatment period.
Time Frame: From first dose of study treatment (Day 1) up to last dose of study treatment, approximately 12 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Caplacizumab and IST Without First-Line TPE
Number analyzed (Participants) | 46
percentage of participants | 2.2 [0.4 to 11.3]

9. Secondary Outcome: Percentage of Participants With Immune-mediated Thrombotic Thrombocytopenic Purpura (iTTP)-Related Death During On-Treatment Period
Description: Percentage of participants with iTTP-related death during on-treatment period are reported.
Time Frame: From first dose of study treatment (Day 1) up to last dose of study treatment, approximately 12 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Caplacizumab and IST Without First-Line TPE
Number analyzed (Participants) | 46
percentage of participants | 0 [0 to 7.7]

10. Secondary Outcome: Percentage of Participants With Immune-mediated Thrombotic Thrombocytopenic Purpura-Related Death During Overall Study Period
Description: Percentage of participants with iTTP-related death during overall study period are reported.
Time Frame: From first dose of study treatment (Day 1) up to end of follow-up (up to approximately 24 weeks)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Caplacizumab and IST Without First-Line TPE
Number analyzed (Participants) | 46
percentage of participants | 0 [0 to 7.7]

11. Secondary Outcome: Percentage of Participants With a Clinical Exacerbation of Immune-Mediated Thrombotic Thrombocytopenic Purpura During On-Treatment Period
Description: Clinical exacerbation was defined as after a clinical response and before a clinical remission, platelet count decreased to <150 × 10^9/L (with other causes of thrombocytopenia excluded), with or without clinical evidence of new or progressive ischemic organ injury, within 30 days of stopping TPE or anti-vWF therapy.
Time Frame: From first dose of study treatment (Day 1) up to last dose of study treatment, approximately 12 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Caplacizumab and IST Without First-Line TPE
Number analyzed (Participants) | 46
percentage of participants | 0 [0 to 7.7]

12. Secondary Outcome: Percentage of Participants With a Clinical Exacerbation of Immune-Mediated Thrombotic Thrombocytopenic Purpura During Overall Study Period
Description: as for outcome 11
Time Frame: From first dose of study treatment (Day 1) up to end of follow-up (up to approximately 24 weeks)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Caplacizumab and IST Without First-Line TPE
Number analyzed (Participants) | 46
percentage of participants | 0 [0 to 7.7]

13. Secondary Outcome: Percentage of Participants With a Clinical Relapse of Immune-Mediated Thrombotic Thrombocytopenic Purpura During On-Treatment Period
Description: Clinical relapse was defined as after a clinical remission, platelet count decreased to <150 × 10^9/L (with other causes of thrombocytopenia ruled out), with or without clinical evidence of new ischemic organ injury. A clinical relapse had to be confirmed by documentation of severe ADAMTS13 deficiency (<10%).
Time Frame: From first dose of study treatment (Day 1) up to last dose of study treatment, approximately 12 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Caplacizumab and IST Without First-Line TPE
Number analyzed (Participants) | 46
percentage of participants | 0 [0 to 7.7]

14. Secondary Outcome: Percentage of Participants With a Clinical Relapse of Immune-Mediated Thrombotic Thrombocytopenic Purpura During Overall Study Period
Description: as for outcome 13
Time Frame: From first dose of study treatment (Day 1) up to end of follow-up (up to approximately 24 weeks)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Caplacizumab and IST Without First-Line TPE
Number analyzed (Participants) | 46
percentage of participants | 0 [0 to 7.7]

ADVERSE EVENTS:
Time Frame: Adverse events collected from first dose of study treatment (Day 1) up to last dose of study treatment + 28 days (approximately 16 weeks). All-cause mortality (death) was assessed from signing of the informed consent form to end of follow-up, approximately 109 weeks.
Description: Analysis was performed on safety population.
Arm/Group | Caplacizumab and IST Without First-Line TPE
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 7/50
Other Adverse Events (participants affected / at risk) | 40/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caplacizumab and IST Without First-Line TPE (N=50)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Anaphylactic Reaction (Immune system disorders) | 1 (1)
Steroid Diabetes (Metabolism and nutrition disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Heavy Menstrual Bleeding (Reproductive system and breast disorders) | 1 (1)
Platelet Count Decreased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caplacizumab and IST Without First-Line TPE (N=50)
Nasopharyngitis (Infections and infestations) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (4)
Steroid Diabetes (Metabolism and nutrition disorders) | 3 (3)
Middle Insomnia (Psychiatric disorders) | 4 (4)
Dizziness (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 18 (21)
Hypoaesthesia (Nervous system disorders) | 3 (3)
Haematoma (Vascular disorders) | 4 (7)
Hypertension (Vascular disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Constipation (Gastrointestinal disorders) | 3 (3)
Gingival Bleeding (Gastrointestinal disorders) | 7 (8)
Petechiae (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Fatigue (General disorders) | 4 (4)
Injection Site Bruising (General disorders) | 4 (4)
Oedema Peripheral (General disorders) | 7 (7)
Pyrexia (General disorders) | 3 (3)
Alanine Aminotransferase Increased (Investigations) | 8 (8)
Blood Bilirubin Increased (Investigations) | 3 (3)
Blood Creatinine Increased (Investigations) | 3 (4)
Troponin Increased (Investigations) | 3 (4)
Contusion (Injury, poisoning and procedural complications) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2024-09-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT05468320/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT05468320/SAP_001.pdf